CLINICAL TRIAL: NCT04691544
Title: Donor Versus Autologous Fecal Microbiota Transplantation for Irritable Bowel Syndrome: a Double Blind, Placebo-Controlled, Randomized Trial
Brief Title: Donor Versus Autologous Fecal Microbiota Transplantation for Irritable Bowel Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Oslo University Hospital (Other); Sorlandet Hospital HF (Other Government); Haukeland University Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 183984
Record Dates: First submitted 2020-12-15; First posted 2020-12-31 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: fecal microbiota therapy; bacteriotherapy; stool transplant; IBS; FMT; gut microbiota brain axis; functional disorder; IBS-M; IBS-D; IBS-C
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Triple blind randomized, placebo controlled, parallell-group multi center trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fecal microbiota transplant from donor A (Active Comparator): One FMT delivered by enema
  Interventions: Biological: Fecal microbiota transplantation (FMT)
- Fecal microbiota transplant from donor B (Active Comparator): One FMT delivered by enema
  Interventions: Biological: Fecal microbiota transplantation (FMT)
- Fecal microbiota transplant from donor C (Active Comparator): One FMT delivered by enema
  Interventions: Biological: Fecal microbiota transplantation (FMT)
- Fecal microbiota transplant from autologous feces (Placebo Comparator): One FMT delivered by enema
  Interventions: Biological: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) — Delivered by enema

SUMMARY:
Many patients with irritable bowel syndrome (IBS) do not experience adequate symptom relief with current treatments. The pathophysiology of IBS is diverse, controversial and not completely understood. The next disruptive frontier would be to find a cure where the effect is predictable and lasting. The study groups phase 2 pilot trial was the first indication of a possible benefit from treating IBS with fecal microbiota transplantation (FMT) (Number needed to treat only five) (Fecal microbiota transplantation versus placebo for moderate-to-severe irritable bowel syndrome: a double-blind, randomized, placebo-controlled, parallel-group, single-centre trial he Lancet Gastroenterology and Hepatology 2018). Additional results from the same trial show that the treatment response may be predicted (unpublished data), and that the pathophysiologic mechanisms behind the treatment response also can be identified (Effects of fecal microbiota transplantation in subjects with irritable bowel syndrome are mirrored by changes in gut microbiome, Gut Microbes 2020). This study is the first phase 3 trial of FMT for IBS worldwide.

The hypothesis of the trial is that donor FMT is more effective than placebo FMT in treating IBS, with little adverse events or complications. Patients ≥18 years with IBS are enrolled at five Norwegian Hospitals in this double blind randomized, placebo controlled, parallell-group multi center trial. Participants are randomized to FMT from a healthy donor (intervention group), or their own feces (placebo group). The primary outcome is the proportion of patients with ≥75 points decrease in the Irritable bowel Symptom Severity score 90 days after treatment.

ELIGIBILITY:
Inclusion

* Diagnosed with IBS in the primary or secondary health care service
* Aged 18-65 years with IBS defined by the Rome IV criteria:
* Moderate to severe IBS symptoms, as defined by a score of ≥175 on the IBS-SSS
* All participants >50 years: Colonoscopy within the last 5 years prior to study entry including negative mucosal biopsy for microscopic colitis in participants subtyped as IBS-D

Exclusion

* Planned evaluations or examinations for bowel related complaints
* Known presence of:

  * Endometriosis or polycystic ovarian syndrome
  * Diabetes type 1 and 2
  * Systemic disease including
* Morbidly obesity (BMI ≥35)
* Severe autoimmune disease
* Severe immune deficiency (acquired, congenital or due to medication)
* Previous treatment with FMT
* History of:

  * Severe psychiatric disorder, alcohol or drug abuse. Mood disorders are allowed as long as there is no reason to believe that it will interfere with the ability to participate in the study.
  * Inflammatory bowel disease, microscopic colitis, diverticulitis or ileus
  * Abdominal surgery, with the exception of appendectomy, cholecystectomy, caesarean section and hysterectomy
  * Malignant disease (excluding basalioma)
* "Red flags'' indicating severe undiagnosed disease including:

  * Night sweats (Repeated episodes of extreme perspiration that may soak nightclothes or bedding)
  * Unintentional weight loss (≥ 4.5 kilograms, or 5% of normal body weight) over less than 12 months without knowing the reason
* Family history of GI cancer defined as two or more first- or second-degree relatives, with:

  * ≥ 1 diagnosed by age 50, OR
  * ≥ 3 first- or second-degree relatives with GI cancer diagnosis, independent of age
* Use of the following the previous 4 weeks:

  * Drugs with effects on bowel function..Rescue medication, such as Polyethylene glycol (Laxabon, Movieprep, Movicol) or Loperamide is allowed
  * Drugs with analgesic action. Use of paracetamol, Non.Steroid Anti-Inflammatory Drugs ≤3 days week is allowed.
* Use of proton pump inhibitors or other antacids ≥3 days week
* Introduction of antidepressants or anxiolytics the last 12 weeks. Patients on a stable dose >12 weeks are eligible.
* Treatment with antibiotics 12 weeks prior to study entry.
* Use of kolestyramin for bile acid malabsorption
* Pregnant, lactating or planning pregnancy.
* Physical exam indicating undiagnosed malignant, autoimmune, or infectious disease
* Laboratory work up indicating undiagnosed digestive, malignant, autoimmune, infectious disease or alternative diagnosis to the IBS related signs and symptoms. The work up includes:

  * Full blood count
  * Erythrocyte sedimentation rate (ESR)
  * C-reactive protein
  * Anti-tissue transglutaminase IgA, total IgA
  * Lactase genotype
  * Stool tests for:
  * Occult blood (Hemofec©).
  * Fecal calprotectin indicating inflammatory bowel disease. The detection limit that excludes participants will depend on which assays is used for analysis at the different study centers.
  * Only if indicated by the patient history (i.e. travelers diarrhea): Stool test for fecal ova and parasite, Clostridoides difficile toxin and pathogenic bacteria (Shigella spp, Salmonella spp. Campylobacter spp, Yersinia spp, and toxin-producing Clostridoides difficile.) All test results must be negative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion in the donorFMT (dFMT) versus autologousFMT (aFMT) group with ≥75 points decrease in the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) day 90 after treatment when compared to the score 8 days before treatment | Day 90 after treatment
  Scores on the IBS-SSS can range from 0 to 500 with higher scores indicating more severe symptoms. The IBS-SSS has five items. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS. A decrease of 50 points is associated with a clinically meaningful improvement.

SECONDARY OUTCOMES:
Proportion in dFMT versus aFMT group with ≥75 points decrease in the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) day 365 after treatment when compared to the score 8 days before treatment | Day 365 after treatment
Proportion of patients in dFMT versus aFMT group with a ≥14 points increase in the IBS-Qualiy of Life (IBS-QoL) day 90 after treatment when compared to the score 8 days before treatment | Day 90 after treatment
  The IBS-QoL is a validated self-report questionnaire specific to IBS to evaluate quality of life over the past 30 days. It consists of 34 items, each with a five-point Likert scale. The individual response to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life. The cut-off for meaningful clinical improvement is set at ≥14 points. There are also eight subscale scores for the IBS-QOL (Dysphoria, Interference with Activity, Body Image, Health Worry, Food Avoidance, Social Reaction, Sexual, Relationships)
Proportion in the dFMT vs aFMT group with 2 or more weeks with treatment success in Adequate relief by the Global Improvement Scale and Abdominal pain day 69, 76, 83 and 90 after treatment. For treatment success criteria A. and B. have to be fulfilled | Day 69, 76, 83 and 90 after treatment
  * A. Adequate relief is determined by the patient question "How would you rate your IBS signs and symptoms overall over the past 7 days?". Criteria A. is fulfilled when participants score 1 or 2 on a 7-point numerical rating scale.
  * B. Abdominal pain is determined by the question "How would you rate your abdominal pain overall over the past 7 days?" The patient answer on a 11-point numerical rating scale, where 0 is "No pain" and 10 is "Worst possible pain''. Criteria B. is fulfilled when participants experience a 30% decrease in the scale score after treatment, compared to the score before treatment.
Proportion of adverse events and serious adverse events in the dFMT versus aFMT group from treatment and until day 90 after treatment | Day 90 after treatment
Proportion of adverse events and serious adverse events in the dFMT versus aFMT group from treatment and until day 90 after treatment | Day 365 after treatment
Change in the dFMT vs aFMT group in mean stool consistency score in the period 8-2 days before treatment, compared to mean stool consistency score in the period 84-90 and 359-365 days after treatment. | 2-8 days before treatment and day 84 to 90 and day 259 to 365 after treatment
  This endpoint only apply to participants subtyped with IBS-diarrhea before treatment.
  Mean stool consistency score is measured by Bristol Stool Scale ("How would you rate the stool consistency overall the last 24 hours?").
  Mean stool consistency score will be derived from: (Sum of each rating by the Bristol Stool Form Scale in a period )/(Number of ratings in a period).
Change in the dFMT vs aFMT group in mean number of complete spontaneous bowel movements (CSBM) in the period 8-2 days before treatment, compared to CSBM in the period 84-90 and 359-365 days after treatment | 2-8 days before treatment and day 84 to 90 and day 259 to 365 after treatment
  This endpoint only apply to participants subtyped with with IBS-constipation before treatment.
  CSBM is measured by the question. "How many CSBM have you passed the last 24 hours?" reported by the participant every second day for eight days?''
  Mean number of complete spontaneous bowel movements will be derived from: (Sum of number of CSBM in each period)/number of assessments of CSBM in a period)
Change in the dFMT vs aFMT group in bowel-related complaints by the item specific and global Irritable Bowel Syndrome Symptom Severity Score score from before and until after treatment. | 8 days before treatment and until 30, 90, 180 and 365 days after treatment
Change in the dFMT vs aFMT group in quality of life by the global and subdomain specific score in the Irritable Bowel Syndrome-Qualiy of Life from before and until after treatment. | 8 days before treatment and until 90, 180 and 365 days after treatment
Change in the dFMT vs aFMT group in fatigue by the global and subdomain specific score in the Modified Fatigue Impact Scale from before and until after treatment. | 8 days before treatment and until 90, 180 and 365 days after treatment
  Items on the MFIS can be aggregated into three subscales (physical (range 0 to 36), cognitive (range 0 to 40), and psychosocial (range 0 to 8)), as well as into a total MFIS score (range 0 to 84). All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.
Change in the dFMT vs aFMT group in anxiety and depression (HADS) by the global and subdomain specific score on the Hospital Anxiety and Depression Scale from before and until after treatment. | 8 days before treatment and until 90, 180 and 365 days after treatment
  The HADS is a fourteen item scale where seven of the items relate to anxiety and seven to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Higher scores indicates higher levels of anxiety or depression
Proportion of participants identified as treatment success (as defined by the primary endpoint) by a ten species profile generated from a metagenomic dataset from the pilot REFIT trial (unpublished data) | Day 90
Change in HRV in donor FMT vs placebo FMT group derived from the R-R intervals in continuous ECG recordings. The primary vagal function outcome will be differences in changes from pre-post treatment between groups in High Frequency HRV (HF-HRV; in ms2). | 90 days after treatment
  Firstbeat Bodyguard will record R-R interval and the Firstbeat life style assessment software will analyze the R-R interval recording and provide the outcome measure
Change in HRV in donor FMT vs placebo FMT group derived from the R-R intervals in continuous ECG recordings. The secondary vagal function outcome will be differences in changes from pre-post treatment between groups in RMSSD (RMSSD; in ms2). | 90 days after treatment
Difference in mean baseline HRV (HF-HRV and RMSSD) between responders' vs non-responders to donor FMT. | 90 days after treatment
  As defined by the primary endpoint in the clinical phase III study, a responder will be defined by a decrease of 75 points from baseline in the irritable bowel symptom severity score 90 days after the intervention with FMT. To determine HRV in each group we will use High Frequency Power analysis denominating HRV in ms2.

OTHER OUTCOMES:
Changes in taxonomy and function of the microbiome, the immune system, metabolome and gut epithelial barrier in participants with vs without treatment success to dFMT and aFMT from before and until after treatment. | 8 days before treatment and until 90 and 365 days after treatment
  This exploratory endpoint will be further specified when all participants has completed their 12 months follow up after treatment. To explore the changes described above stool, serum, plasma and urine is obtained from participants before and at 90 and 365 days after treatment. The biobanking at 365 will only be performed on a subset of participants. Stool from each donor feces donation will also be biobanked.
Differences in taxonomy and function of the microbiome, the immune system, metabolome and gut epithelial barrier before treatment in FMT donors vs participants with vs without treatment success to dFMT and aFMT from before and until after treatment. | 8 days before treatment and until 90 and 365 days after treatment
  This exploratory endpoint will be further specified when all participants has completed their 12 months follow up after treatment. To explore the changes described above stool, serum, plasma and urine is obtained from participants before and at 90 and 365 days after treatment. The biobanking at 365 will only be performed on a subset of participants. Stool from each donor feces donation will also be biobanked.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Johnsen, MD PhD, Principal Investigator — Univeristy Hospital of North Norway; Rasmus Goll, MD PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- Ålesund Hospital, Ålesund, Norway